CLINICAL TRIAL: NCT01734642
Title: A Regional Project to Reduce Adverse Drug Reactions Due to Medication Errors in Hospital
Brief Title: Observational Study to Reduce Medication Errors
Acronym: OSME
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Universita di Verona (Other)
Collaborators: Ospedale S.Bortolo -Vicenza, Italy (Unknown); Ospedale Mater Salutis-Legnago(Verona), Italy (Unknown); Ospedale Fra Castoro- San Bonifacio (Verona), Italy (Unknown); Azienda Ospedaliera Universitaria Integrata Verona (Other)
Responsible Party: Principal Investigator, GIAMPAOLO VELO, Prof. of Pharmacology and Director of the Clinical Pharmacology Unit, Verona, Italy, Universita di Verona
Other Study IDs: 31025
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2012-11-29 (Estimated); Status verified 2012-11

CONDITIONS: Medication Errors
Keywords: Medication errors, patients hospitalized, ADRs, adverse events

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- PATIENT HOSPITALIZED: ALL THE PATIENTS HOSPITALIZED IN THE INVOLVED UNITS WHO GAVE THEIR INFORMED CONSENT. PATIENTS HOSPITALIZED DURING THE WEEK-END WILL BE ENROLLED ON the next MONDAY

SUMMARY:
A medication error is a failure in the treatment process that leads to, or has the potential to lead, to harm to the patient.1 Medication errors are a common unfortunate occurrence in hospital. They can occur in different phases of the therapeutic process (prescribing, distribution, administration and monitoring) and have significant impact on morbidity and mortality. Prescribing faults and prescription errors are major problem among medication errors .Prescription errors account for 70 % of medication errors that could potentially result in adverse drug effects.2 Overall it has been estimated prescription errors affect 7 % of medication orders, 2% of patient days and 50 % of hospital admissions.3,4 When harm arises from a medication error it is potentially preventable. The medication errors project was devised to analyze and limit through educational audit and other tools, as much as possible, damages due to the therapeutic process. The project will include 5 phases. Preliminary phase: organizational meetings. Phase I: Patient monitoring: a monitor in collaboration with health professionals of involved units will review all patient charts and will register all adverse drug reactions(ADRs). All ADRs will be introduced by the monitor in a database. Health professional will be invited to send the reports of observed ADRs. Evaluation of ADRs : a panel of experts will evaluate if the ADRs are due to medication errors or not. Phase II :educational audits directed to health professionals will be organized. Tools to reduce the medication errors will be proposed. Phase III: the same procedure of the first phase. Final phase (IV): analysis of data with publication of a scientific article.

ELIGIBILITY:
Inclusion Criteria:

* all patients hospitalized in the involved units who gave their informed consent. Patients hospitalized during the week-end will be enrolled on the next monday.

Exclusion Criteria:

* all patients with evident mental and physical problems and all patients who did not give their informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients from 18 to 65 and over 65 years old hospitalized in the involved departments during the study period.
Sampling Method: Probability Sample
Enrollment: 8000 (Estimated)
Dates: Start 2013-01; Primary Completion 2013-11 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse drug reactions due to medication errors occurring during hospitalization | within the first 3 months

SECONDARY OUTCOMES:
Number of participants with preventable ADRs due to medication errors | 3 months

OTHER OUTCOMES:
the impact of educational audit will be evaluated | during the final phase

CONTACTS AND LOCATIONS:
Overall Officials: Giampaolo Velo, Medicine and Surgery, Study Director — The University of Verona, Verona , Italy
Locations (4):
- Italy (4):
  - Mater Salutis Hospital, Legnago, Verona
  - Fracastoro Hospital, San Bonifacio, Verona
  - University Hospital of Verona (AOUI), Verona, Italy, Verona, Verona
  - San Bortolo Hospital, Vicenza, Vicenza

REFERENCES:
- [Background] Aronson JK. Medication errors: definitions and classification. Br J Clin Pharmacol. 2009 Jun;67(6):599-604. doi: 10.1111/j.1365-2125.2009.03415.x. PMID 19594526
- [Background] Velo GP, Minuz P. Medication errors: prescribing faults and prescription errors. Br J Clin Pharmacol. 2009 Jun;67(6):624-8. doi: 10.1111/j.1365-2125.2009.03425.x. PMID 19594530
- [Background] Bates DW, Teich JM, Lee J, Seger D, Kuperman GJ, Ma'Luf N, Boyle D, Leape L. The impact of computerized physician order entry on medication error prevention. J Am Med Inform Assoc. 1999 Jul-Aug;6(4):313-21. doi: 10.1136/jamia.1999.00660313. PMID 10428004
- [Background] Lewis PJ, Dornan T, Taylor D, Tully MP, Wass V, Ashcroft DM. Prevalence, incidence and nature of prescribing errors in hospital inpatients: a systematic review. Drug Saf. 2009;32(5):379-89. doi: 10.2165/00002018-200932050-00002. PMID 19419233